

#### **RESEARCH PROPOSAL**

#### TITLE:

# THE FEASIBILITY AND IMPACT OF A HOME-BASED NMES PROGRAM ON POST-STROKE LOWER LIMB SPASTICITY

Principle investigator : Dr. Raja Nabila binti Raja Mohamed Anuar

Department of Rehabilitation Medicine, University of Malaya

Medical Centre

Supervisor : Dr Chung Tze Yang

Department of Rehabilitation Medicine, University of Malaya

**Medical Centre** 

Co-investigators : 1. Pn Ida Mardiana binti Mohamad Yusop

Physiotherapy Division, Department of Rehabilitation Medicine,

University of Malaya Medical Centre

2. Pn Wahida binti Wahid

Physiotherapy Division, Department of Rehabilitation Medicine,

University of Malaya Medical Centre

Study site : University of Malaya Medical Centre (UMMC)

Version : 1.0

Date : 1<sup>st</sup> April 2020

Time Frame : 1<sup>st</sup> July 2020 – 30<sup>th</sup> September 2021

## **CONTENTS**

| No | Торіс | Page |
|---|---|---|
| 1 | LIST OF ABBBREVIATIONS | 3 |
| 2 | ABSTRACT | 4 |
| 3 | INTRODUCTION 3.1 Research Area 3.2 Research Questions 3.3 Objectives 3.4 Significance of study | 5<br>5<br>5<br>6 |
| 4 | LITERATURE REVIEW | 6 |
| 5 | METHODOLOGY 5.1 Study Design 5.2 Setting 5.3 Study Population 5.4 Inclusion Criteria 5.5 Exclusion Criteria 5.6 Intervention, dose and mode of administration 5.7 Outcome measures 5.8 Sample Size 5.9 Study Flow Chart 5.10 Data Analysis | 10<br>10<br>10<br>10<br>10<br>11<br>11<br>11<br>12<br>12 |
| 6 | STRENGTH AND LIMITATIONS | 13 |
| 7 | TIMELINE | 13 |
| 8 | REFERENCES | 14 |
| 9 | APPENDIX | 16 |

## 1. LIST OF ABBREVIATIONS

| PSS | Poststroke spasticity |
|------|----------------------------------------|
| UMMC | University of Malaya Medical Centre |
| NMES | Neuromuscular Electrical Stimulation |
| MAS | Modified Ashworth Scale |
| QoL | Quality of Life |
| PF | Plantarflexors |
| DF | Dorsiflexor |
| PC | Pulsed Current |
| PD | Pulse Duration |
| Hz | Hertz |
| s | second |
| mcs | Microseconds |
| SPSS | Statistical Package For Social Science |

#### 2. ABSTRACT

**BACKGROUND:** Spasticity is a common complication post stroke. Post-stroke spasticity along with weakness and lack of coordination result in gait abnormalities and problems with upper limb function. This affects stroke survival negatively on health-related QoL, affecting the caregiver and is a socioeconomic burden. Treatment options of spasticity includes physical therapy, ankle-foot orthosis, oral medications; chemodenervation with botulinum toxins, phenol, or alcohol; intrathecal baclofen, and surgical interventions. Recent treatment options include neuromuscular electric stimulation (NMES), a form of therapy that applies electrical currents to produce contraction of innervated muscle by depolarizing local motor nerves. Currently, there are wide varieties of devices delivering NMES, including battery-operated, portable devices. The purpose of this study is to evaluate the feasibility and acceptability of homebased NMES program on lower limb spasticity following stroke. We also like to assess the impact of the program to lower limb spasticity. To date there is no such research available in Malaysia.

#### **OBJECTIVES:**

- 1. To evaluate the feasibility and acceptability of home based NMES program.
- 2. To assess the impact of home based NMES program in post stroke spasticity (spastic ankle plantarflexors)

METHOD: Single arm prospective cohort intervention study. Participants are patients (post stroke >6months) with ankle plantarflexors spasticity Modified Ashworth Scale (MAS) 1+ to 3. Patient will receive homebased NMES for 20minutes, 5days a week for 4 weeks with stretching exercises while they resume their usual conventional rehabilitation program. NMES dose: Biphasic pulsed current, 50Hz, pulse width 400μs, ON:OFF 10:20s with amplitude individual maximum tolerated to achieve ankle dorsiflexion, with electrodes at common peroneal nerve and motor point of tibialis anterior muscle. Patient will receive NMES treatment in sitting position with sole contact with the floor. Feasibility is determined by retention and compliance rates; acceptability by structured questionnaire at the end of study and the impact is determined by outcome measure of plantarflexors MAS, Modified Tardieu Scale, dorsiflexor strength and 10 meter walking test.

#### 3. INTRODUCTION

#### 3. 1 Research Area

Spasticity is a common complication post stroke. The prevalence of spasticity ranging from 19% at 3 months post stroke to 46% at 12 months post stroke. <sup>1-3</sup> Spasticity is defined as "a motor disorder characterized by a velocity-dependent increase in tonic stretch reflexes with exaggerated tendon jerks, resulting from hyperexcitability of the stretch reflex, as one component of the upper motor neuron syndrome". <sup>4</sup> The impact of post stroke spasticity is substantial. Post-stroke spasticity along with weakness and lack of coordination, affects stroke survival negatively on the gait, functional activity and on the health-related quality of life (QoL). It also affects the caregiver on their QoL as increased care that the stroke survivor with spasticity requires, and it is a socioeconomic burden. <sup>5</sup> A study in Sweden reported 4-fold increase in direct costs for patients with stroke with spasticity compared with patients with stroke without spasticity. <sup>6</sup>

There are a number of treatment options for management of spasticity, including physical therapy; the usage of ankle-foot orthosis (AFO), oral medications; chemodenervation with botulinum toxins (BoNT), phenol, or alcohol; intrathecal baclofen therapy; and surgical interventions. <sup>7,8</sup> More recent treatment options include neuromuscular electric stimulation (NMES). <sup>7–9</sup> NMES refers to forms of therapy that apply electrical currents to produce contraction of innervated muscle by depolarizing local motor nerves. Currently there are wide variety of devices deliver NMES, including battery-operated, portable devices <sup>10</sup>. However, NMES as a treatment of spasticity is not widely used in our local population. The purpose of this study is to evaluate the feasibility and acceptability of homebased NMES program on lower limb spasticity following stroke. We also like to assess the impact of the program to lower limb spasticity. To date there is no such research available in Malaysia.

#### 3.2 Research Questions

- 1. Does home based NMES program is feasible and acceptable for patient with post stroke spasticity?
- 2. Does home based NMES improve post-stroke spasticity of lower extremities (spastic ankle plantarflexors) assessed clinically and functionally (Modified Ashworth Scale (MAS), Modified Tardieu Scale and walking speed)?

#### 3.3 Objective

- 1. To evaluate the feasibility and acceptability of home based NMES program in post-stroke patient with spasticity.
- 2. To assess the impact of home based NMES program in lower limb spasticity (spastic ankle plantarflexors) following stroke in direct clinical measurement and functionally.

#### 3.4 Significance of this study

- 1. This is first study in Malaysia that utilizes NMES for lower limb spasticity. The NMES devices are easily available commercially and relatively cheap. By conducting this study, we can assess the feasibility and patient's perceptions of home-based NMES program for post-stroke population and will assist us in further prescription and management of post-stroke patient.
- 2. It is homebased program. Formulating home-based rehabilitation protocol is substantial for rehabilitation medicine to provide better accessibility, maximize participation and empower patient-driven rehabilitation. Furthermore, with current trend (eg pandemic, logistic issue etc) patient preferred for less frequent hospital visitation; hence strengthening of home-based program is crucial. Thus, we can maintain rehab efficacy with reduced hospital visit and home program.
- 3. The result of this study will give us further knowledge on the usage of NMES and spasticity management. It enables healthcare professionals to decide on management of spasticity which is possibly less invasive, safe and more cost efficient.

#### 4.0 Literature review

| N | Title, Author, year | Type of study, sample size, Population and Methodology | NMES parameters and outcome measures | Result |
|---|---|---|---|---|
| 1. | The feasibility | Single arm prospective | Frequency: 50 Hz, | The results of the pilot |
| | and acceptability | pilot study | PD: 300 mcs | study suggest that |
| | of neuromuscular | N 15-> 10(completed) | On/off: 5s on 5 s off | NMES is both feasible |
| | electrical | | intensity was individually to | and acceptable in a |
| | stimulation to | Intervention: daily NMES | obtain tetanic contraction or | mixed group of |
| | improve exercise | at quadriceps | maximum tolerated intensity | patients with cancer, |
| | performance in | | | most of whom had |
| | patients with | Objectives: | 30min/d, 6 weeks | poor performance |
| | advanced cancer: | 1) to evaluate the | | status. |
| | a pilot study <sup>11</sup> | acceptability and | Placement: at vastus medialis | |
| | | feasibility of a home | oblique distally, | Does not demonstrate |
| | Tamara Windholz, | based NMES | midpoint of quadriceps mm | that NMES leads to |
| | Tara Swanson, | intervention in a patients | belly at proximal | improved physical |
| | Brandy L | attending the Cancer | | functioning in cancer |
| | Vanderbyl and R | Nutrition-Rehabilitation | Outcome assessment | patients with poor |
| | Thomas Jagoe. | Program | 1. Feasibility - proportion of pt | performance status, |
| | | clinic at the Jewish | who completed 6/52 | may be due to marked |
| | BMC Palliative | General Hospital (CNR- | intervention, and overall level | heterogeneity in terms |
| | Care 2014 | JGH) | of adherence (40% cut-off) | of medical status and |
| | | | 2. Acceptability NMES | physical functioning; |
| | | 2) To assess the impact | evaluated at the end of 6 weeks | and small sample. |
| | | of the NMES | by questionnaire. | |
| | | intervention on test of | 3. Physical performance | |
| | | physical function. | measures at baseline and at the | |
| | | | end (PS, 6MWT, STC) | |
| 2. | Feasibility of | Prospective cohort study | NMES session for 20min during | Critically ill patients |
| | neuromuscular | (N 50) | 5 days per week + standard PT | having sepsis, edema, |
| | electrical | / | during the stay (positioning, | or receiving |
| | stimulation in | To investigate the | chest PT, ROM and cycling in | vasopressors were less |
| | critically ill | feasibility of NMES in | bed according to pt) | likely to respond to |
| | patients <sup>12</sup> | eliciting a muscle | 0 1 7 | NMES with an |

| | Johan Segers, PT, MSc a, Greet Hermans, MD, PhD b, Frans Bruyninckx, MD, PhD c, Geert Meyfroidt, MD, PhD d, Daniel Langer, PT, PhD a, Rik Gosselink, PT, PhD a Journal of Critical care, 2014 | contraction of the QF in critically ill patients and safety. | NMES session is given in slowly increasing intensitiy and pulse duration in graded fashion to achieve favourable contraction (maximal 80mA and 500 mcs) Outcome measure: 1) Feasibility> Assessing responder (contraction 4-5) or non responder (contraction 1-3) and the factors affecting it: i- level of consciousness ii- Level of edema iii- Sepsis iv-medications 2) Safety: cardioresp response (HR, BP, O2Sat, breathing) skin response | adequate quadriceps contraction. Neuromuscular electrical stimulation is a safe intervention to be administered in the ICU. |
|---|---|---|---|---|
| 3. | Does electrical stimulation reduce spasticity after stroke? A randomized controlled study <sup>13</sup> Amir H Bakhtiary and Elham Fatemy Clinical Rehabilitation, 2008 | RCT N 40 (20 intervention, 20 control) 1) Bobath + NMES 2) Control: Bobath Patient with ankle plantarflexor spasticity (does not mention duration post stroke) | Faradic type PC Frequency 100Hz pulse stimulation PD: 100mcs, On:off 4:6, no ramp time supramaximal (25% over the intensity needed to produce maximum contraction of muscle) 9 minutes daily For 20 session Electrodes: cathode on the tibialis anterior muscle via and anode over the fibula head Outcome measures: 1) Passive ankle joint DF range of motion, 2) DF strength test, 3) PF muscle tone by Modified Ashworth Scale (MAS) 4) soleus muscle H-reflex. | Improvement were greater in treatment group: 1) Lower PF spasticity (MAS) in combination group - 1.6 versus - 1.1 in the Bobath group 2) Higher ankle DF ROM in the combination group Vs in the Bobath group = 11.4 vs 6.1 3) Higher DF strength in combination group (0.7 vs 0.4) |
| 4. | Functional electrical stimulation of dorsiflexor muscle: Effects on dorsiflexor strength, plantarflexor spasticity, and motor recovery | Prospective interventional study. N 51 (27 intervention, 24 control) 1) Conventional rehab program (CRP) + EMS 2) CRP only | Waveform NR Frequency 35Hz PD 280 mcs Stimulation timed to the gait cycle by using a heel switch placed in the shoe, causes ankle dorsiflexion in the swing phase of gait) | Therapy combining EMS and conventional rehabilitation program was superior to a conventional rehabilitation program alone, in terms of: 1) reducing spasticity, - 1.1 vs - 0.5 |

| | in stroke patients <sup>14</sup> Sukanta K. Sabut , Chhanda Sikdar , Ratnesh Kumar and Manjunatha Mahadevappa NeuroRehabilitati on, IOP Press 2011 | >3months post stroke with hemiplegia (unilateral drop foot) and able to walk at least 10m without assistance. Not contracted. | Amplitude set to produce muscle contraction within patient's comfort. Duration: 20–30min 5 days a week, for 12 weeks. Electrode: common peroneal nerve as it passes over the head of the fibula and the motor point of tibialis anterior. Outcome measures: 1) PF spasticity measured by MAS 2) DF strength 3) Active/passive ankle joint dorsiflexion ROM 4) Lower-extremity motor recovery by FMA scale. @0 and week 12. | 2) improving DF ROM and strength 3) lower extremity motor recovery in stroke patients. |
|---|---|---|---|---|
| 5. | The effects of neuromuscular electrical stimulation on clinical improvement in hemiplegic lower extremity rehabilitation in chronic stroke: A single-blind, randomized, controlled trial 15 Nilgun Mesci, Ferda Ozdemir, Derya Demirbag Kabayel & Burcu Tokuc Disability and Rehabilitation 2009 | RCT N 40 (20 intervention, 20 control) Intervention: inpatient CRP + NMES Control: inpatient CRP Hemiparesis due to stroke >3 months, mobility of ankle to permit at least neutral position, MAS <4 | Biphasic PC wave Frequency 50 Hz Pulse width 400 mcs On:off: NR Intensity: fully contracted muscle without discomfort or pain. Duration 20min 5 days, 4 weeks Pt position: sitting position and to keep their soles of their feet in contact with the floor. Electrode: positive active electrode right below the fibular head where the peroneal nerve is going through; and the negative electrode was positioned on the midpoint of the tibialis anterior muscle on the front side of the leg. Outcome measures: 1. Ankle passive DF ROM 2. Spasticity MAS 3. Neurophysiological improvement in the lower extremities in Brunnstrom Stage (BS) 4. Functional Independence Measurement (FIM). | Improvement were greater in treatment group in all outcome measures. 1) ankle DF ROM (6.25 vs 1.0) p=0.000 2) decrease in the MAS -1.2 vs -0.15 (P=0.000) 3) increase in the lower extremity BS 0.8 vs 0.25 (p=0.005) 4) improvement in the Rivermead leg and trunk scores p= 0.004) improvement in the FIM motor subscore (p=0.018) |

| 5. Rivermead Motor | |
|---|---|
| Assessment Scale | |
| 6. Functional Ambulation | |
| Categories (FAC) | |
| 6. Transcutaneous single-blinded, stratified, Square PC Both TE | ENS (TENS and |
| | RT) groups |
| | d earlier and |
| , , , , , | antly greater of<br>on in PF |
| | ity as measured |
| Improves Lower (1) TENS, Duration: 60minutes at week | <b>&lt;</b> 2 |
| Limb Functions in (2) TENS +TRT, 5 days a week for 4 weeks. | |
| | ning TENS with proved outcome |
| | es significantly |
| , | nan TENS alone, |
| PhD; Christina 1 year post stroke and points PLBO+1 W.Y. Hui-Chan, able to walk 10 m treatments | TRT, or no |
| PhD unassisted with or Outcome measurements: | CIII. |
| without walking aids, 1) Composite Spasticity Scale, Improv | ements can |
| Coope of at least 10 and I down they are and plantaged according | e maintained 4 |
| more in their ankle PF recorded with a load cell ended | after treatment |
| (moderate spasticity) mounted on a custom- built | |
| foot frame 2) gait vologity (CALTRita) | |
| 3) gait velocity (GAITRite) | |
| @ baseline, after 2 and 4 weeks | |
| of treatment, and 4 weeks after treatment ended | |
| treatment ended | |
| | review, the |
| | of NMES with a ncy between 30 |
| | Hz and a pulse |
| After Stroke trials were included with extracted was range of motion, width be | etween 0.1 and |
| | for 30 minutes |
| | per week for 3<br>eks were |
| | ted with |
| Controlled Trials <sup>9</sup> success | ful results. |
| Cinara Stein, MSc; | |
| Carolina Gassen | |
| Fritsch, Ft; | |
| Caroline Rebisson MSs: | |
| Robinson, MSc; Graciele Sbruzzi, | |
| DSc; Rodrigo | |
| Della Méa Plentz, | |
| DSc | |
| American Heart | |
| Association, 2015 | |

#### 5. Methodology:

#### 5.1 Study Design

Single arm prospective cohort intervention study. Patient with PSS recruited and will apply NMES to the lower limb at home in addition to their daily stretching exercises of their plantarflexion. They may also resume their conventional outpatient therapy session.

#### 5.2 Setting

- Recruitment: Specialist clinic and therapy areas of Department of Rehabilitation Medicine, UMMC.
- · Intervention: Home setting

#### 5.3 Study population

- Participants who are attending Rehabilitation Medicine Specialist clinics and therapy areas that fulfill the criteria will be screen for eligibility and recruited.
- Demographics of participants including age, sex, race, dominant hand, etiology of stroke (ischemic/hemorrhagic), side of hemiparesis will be recorded.

#### 5.4 Inclusion criteria includes:

- Post stroke (hemorrhagic or ischemic) with ankle plantarflexor (gastrocnemius and soleus)
   spasticity MAS 1+ to MAS 3
- Post stroke more than 6 months
- > 18 years old
- Able to ambulate 10 meter either independently or aided (single point stick or quadripod)
- Compliant to outpatient therapy.
- Minimal cognitive (MMSE> 24) and minimal sensory impairment
- Stable neurological and medical condition

#### 5.5 Exclusion criteria

- Introduction or changes in anti-spastic medication dose within 3 months or during study period
- Receiving intervention for spasticity (eg BoNT or serial casting) within 3 months or during research period.
- New neurological condition/disease
- Presence of contraindications to NMES, which is<sup>17</sup>:
  - Pregnancy
  - Malignancy
  - Presence of electronic implant eg cardiac pacemaker, cardioverter defibrillator
  - Uncontrolled seizure/epilepsy
  - Infected tissues/ tuberculosis or osteomyelitis
  - Impaired lower limb circulation/ DVT/ thrombophlebitis

- Recent fracture or osteoporosis
- Actively bleeding tissue or person with untreated hemorrhagic disorder
- Damaged or skin diseases at the affected lower limb

#### 5.6 Sample Size

Consistent with the feasibility design, no formal sample size calculation was undertaken; rather a target sample of 20 participant was deemed sufficient to provide preliminary data required to test our feasibility study aim.

Furthermore from literature review, Bakhtiary et al reported improvement of plantarflexor spasticity (MAS) in intervention group - 1.6 (SD 0.5) versus - 1.1 (SD 0.31) in control group. Thus the effect size is 0.75, and for an alpha of 0.05 and power of 0.8, sample size of 23 each arm is needed (not considering the attrition rate).

#### 5.7 Intervention, dose and mode of administration<sup>15</sup>:

- It is a home-based NMES applications over the lower limb with plantarflexor spasticity using a commercially available consumer NMES machine.
- Each patient will get a pair of new electrodes.
- Dose of NMSE:
  - NMES waveform: biphasic PC
  - Frequency 50Hz, pulse width: 400μs, ON:OFF 10s:20s
  - Current amplitude: individual maximum tolerated to achieve ankle dorsiflexion.
- Electrode placement (transcutaneous surface electrode):
  - 1 electrode over the common peroneal nerve outlet (below the fibular head),
  - 1 electrode over motor point of tibialis anterior or both tibialis anterior and peronei muscle.
- Body and limb position: Patient sitting with the sole in contact with the floor, and try for active dorsiflexion during stimulation.
- Duration: 20 minutes per session daily, 5 days a week, for 4 weeks (total 20sessions)
- Compliant is monitored by daily logbook (Appendix 1)

#### 5.8 Outcome measures

- Primary Outcome:
  - 1) Feasibility as assessed by proportion of patients who completed the program, and overall level of compliant (retention and compliance rates)
  - 2) Acceptability as evaluated at the end of the intervention by brief structured

questionnaire developed for this study using 5 point Likert scale (Appendix 2)

- Secondary Outcome:
  - 1) Clinical measurement of spasticity and functional outcomes:
    - a. Modified Ashworth Scale (MAS)
    - b. Modified Tardieu Scale (R1 R2 of ankle dorsiflexion)
    - c. Ankle dorsiflexion muscle strength
    - d. 10 meter walking test

#### **5.9 Study Flow Chart**

1) Screening - Inclusion/exclusion criteria application to patients attending Rehabilitation Medicine Specialist clinic and therapist area



2) Consent - Explanation of study, Patient Information Sheet and Written Consent



- 3) Pre-intervention assessment and familiarization session
  - Pre-intervention assessment per outcome measures (MAS, Modified Tradieu Scale, strength, and 10MWT)
  - Teaching patient (with or without family member) application of NMES
  - Trial of a 20 minutes session



- 4) Intervention: Home-based NMES program for 4 weeks
  - A NMES device will be loaned to patient throughout the study period
  - A new pair of self-adhesive electrodes will be given to patient
  - Pre-setting NMES dose: Frequency 50Hz, pulse width: 400μs, ON:OFF 10s:20s
  - daily logbook



- 5) Completion of intervention
  - Submission of logbook and NMES machine
  - post intervention assessment as per outcome measures (MAS, Modified Tradieu Scale, strength, and 10MWT)
  - Post intervention questionnaire

#### 5.10 Data Analysis

Data from this study will be analyzed using Statistical Package for Social Science (SPSS) software.

- Comparison between participants who did and did not complete the study and the compliance rate will be performed using unpaired t-test and Fisher's exact test for continuous and categorical variables respectively.
- Improvement spasticity MAS (grading) paired t-test
- Improvement in ankle dorsiflexion ROM (degree) paired t-test
- Ankle dorsiflexion muscle strength (grading) paired T-test
- 10 meter walking speed (ms-1) paired t-test

#### 6.0 Strength and Limitation

#### Strength

- No previous published study in Malaysia looking at NMES application for reducing spasticity post- stroke.
- Easily available equipment commercially and relatively cheap and safe.
- Study conducted in stroke population therefore adequate number of samples can be recruited.

#### Limitation

- Resource and funding; it will be self-funded by main investigators.
- Equipment handling and maintenance; risk of faulty equipment which could limit the research progress.
- Single centre study

#### 7.0 Timeline

#### **Gantt Chart**



#### 8.0 References

- 1. Sommerfeld DK, Eek EUB, Svensson AK, Holmqvist LW, Von Arbin MH. Spasticity after Stroke: Its Occurrence and Association with Motor Impairments and Activity Limitations. *Stroke*. 2004;35(1):134-139. doi:10.1161/01.STR.0000105386.05173.5E
- 2. Watkins CL, Leathley MJ, Gregson JM, Moore AP, Smith TL, Sharma AK. Prevalence of spasticity post stroke. *Clin Rehabil*. 2002;16(5):515-522. doi:10.1191/0269215502cr512oa
- Article CME. Upper-Limb Spasticity During the First Year After Stroke. 2014;93(10):884-896. doi:10.1097/PHM.000000000000157
- 4. Feldman, young K. Lance JW. Symposium Synopsis. In: Feldman RG, Young R, Koella WP, Eds. Spasticity: Disordered Motor Control. Chicago, IL: Year Book Medical Publishers; 1980:485–494.; 1980.
- 5. Zorowitz RD, Gillard PJ, Brainin M. Poststroke spasticity: Sequelae and burden on stroke survivors and caregivers. *Neurology*. 2013;80(3 SUPPL.2). doi:10.1212/wnl.0b013e3182764c86
- 6. Lundström E, Smits A, Borg J, Terént A. Four-fold increase in direct costs of stroke survivors with spasticity compared with stroke survivors without spasticity: The first year after the event. *Stroke*. 2010;41(2):319-324. doi:10.1161/STROKEAHA.109.558619
- 7. Francisco GE, McGuire JR. Poststroke spasticity management. *Stroke*. 2012;43(11):3132-3136. doi:10.1161/STROKEAHA.111.639831
- 8. Jacob A, Wilkenfeld L. Review of electrical stimulation, botulinum toxin, and their combination for spastic drop foot. 2013;50(3):315-326.
- 9. Stein C, Fritsch CG asse., Robinson C, Sbruzzi G, Plentz RD ell. M. Effects of Electrical Stimulation in Spastic Muscles After Stroke: Systematic Review and Meta-Analysis of Randomized Controlled Trials. *Stroke*. 2015;46(8):2197-2205. doi:10.1161/STROKEAHA.115.009633
- 10. Nussbaum EL, Houghton P, Anthony J, Rennie S, Shay BL, Hoens AM. Neuromuscular electrical stimulation for treatment of muscle impairment: Critical review and recommendations for clinical practice. *Physiother Canada*. 2017;69(5 Special Issue):1-76. doi:10.3138/ptc.2015-88
- 11. Windholz T, Swanson T, Vanderbyl BL, Jagoe RT. Erratum: The feasibility and acceptability of neuromuscular electrical stimulation to improve exercise performance in patients with advanced cancer: A pilot study (BMC Palliative Care (2014) 13 (33)). *BMC Palliat Care*. 2014;13(1):1-8. doi:10.1186/1472-684X-13-33
- 12. Segers J, Hermans G, Bruyninckx F, Meyfroidt G, Langer D, Gosselink R. Feasibility of neuromuscular electrical stimulation in critically ill patients. *J Crit Care*. 2014;29(6):1082-1088. doi:10.1016/j.jcrc.2014.06.024
- 13. Bakhtiary AH, Fatemy E. Does electrical stimulation reduce spasticity after stroke? A randomized controlled study. *Clin Rehabil*. 2008;22(5):418-425. doi:10.1177/0269215507084008
- 14. Sabut SK, Sikdar C, Kumar R, Mahadevappa M. Functional electrical stimulation of dorsiflexor muscle: Effects on dorsiflexor strength, plantarflexor spasticity, and motor recovery in stroke patients. NeuroRehabilitation. 2011;29(4):393-400. doi:10.3233/NRE-2011-0717
- 15. Mesci N, Ozdemir F, Kabayel DD, Tokuc B. The effects of neuromuscular electrical stimulation on clinical improvement in hemiplegic lower extremity rehabilitation in chronic stroke: A single-blind, randomised, controlled trial. *Disabil Rehabil*. 2009;31(24):2047-2054. doi:10.3109/09638280902893626
- 16. Ng SSM, Hui-Chan CWY. Transcutaneous electrical nerve stimulation combined with task-related training improves lower limb functions in subjects with chronic stroke. *Stroke*. 2007;38(11):2953-2959. doi:10.1161/STROKEAHA.107.490318

- 17. Rennie S. *ELECTROPHYSICAL AGENTS Contraindications And Precautions: An Evidence-Based Approach To Clinical Decision Making In Physical Therapy.* Vol 62.; 2010. doi:10.3138/ptc.62.5
- 18. Kondo T, Yamada S, Tanimura D, et al. Neuromuscular electrical stimulation is feasible in patients with acute heart failure. *ESC Hear Fail*. 2019;6(5):975-982. doi:10.1002/ehf2.12504

# Appendix 1

#### Patient's Feedback Questionnaire

| | | | | | illali e | | Date: | | |
|---|---|---|---|---|---|---|---|---|---|
| | General acceptability and satisfaction | | 1=<br>Stror | | 2 =<br>Disa | gree | 3 =<br>Neutral | 4 =<br>Agree | 5 =<br>Strongly<br>Agree |
| 1. | Using the NMES for 4 weeks is acceptable | | | | | | | | |
| 2. | Using NMES for 20 minutes a day is acceptable | | | | | | | | |
| 3 | Using NMES had a positive impact on my lower limb spasticity | | | | | | | | |
| 4. | Using NMES had a positive impact on my ambulation | | | | | | | | |
| 5. | I would continue/repeat the NMES program after the study | er | | | | | | | |
| 6. | I would recommend this program to my colleagues/other patients | | | | | | | | |
| 7 | Overall, I think the homebased NMES program is good intervention | s a | | | | | | | |
| 8. | I would consider buying the device if the price is affordable | | | | | | | | |
| | Device's operation experiences. | | 1=<br>Strong<br>Disagr | - | 2 =<br>Disag | ree | 3 =<br>Neutral | 4 =<br>Agree | 5 =<br>Strongly<br>Agree |
| 9. | The NMES device is simple to use | | | | | | | | |
| 10. | Most of the time I can handle the device independently. | | | | | | | | |
| 11. | It is easy to put on the surface electrode to the lower limb. | | | | | | | | |
| 15. | I can use the surface electrode independently | | | | | | | | |
| | While using the NMES, I have experience | 1:<br>N | =<br>ever | 2 =<br>Rai | rely | 3 =<br>Son | netimes | 4 =<br>Often | 5 =<br>Always |
| 16 | Pain | | | | | | | | |
| 17 | Discomfort | | | | | | | | |
| 18 | Skin irritations/ burns | | | | | | | | |
| | Muscle fatigue | | | | | | | | |
| 19 | | | | | | | | | |

# Appendix 2

## **HOME-BASED NMES PROGRAM LOG SHEET**

| No Date Time start Time end NMES intensity Stretching Notes | Na | me: | | | | | |
|---|---|---|---|---|---|---|---|
| Week 1: No Date Time start Time end NMES intensity Stretching Notes 1. | RN | I/ IC: | | | | | |
| No Date Time start Time end NMES intensity Stretching Notes | Per | riod: | to | | | | |
| No Date Time start Time end NMES intensity Stretching Notes | | | | | | | |
| 1. | We | eek 1: | | | | | |
| 2. | No | Date | Time start | Time end | NMES intensity | Stretching | Notes |
| 4. | 1. | | | | | | |
| 4. | 2. | | | | | | |
| Outpatient therapy session: Yes/ No Date: Time: From | 3. | | | | | | |
| Outpatient therapy session: Yes/ No Date: Time: From | 4. | | | | | | |
| Date: Time: Fromto Place: Week 2 No Date Time start Time end NMES intensity Stretching Notes | 5. | | | | | | |
| Date: Time: Fromto Place: Week 2 No Date Time start Time end NMES intensity Stretching Notes | | | | | | | |
| 1. | Dat<br>Tim<br>Pla | te:<br>ne: From<br>nce:<br>eek 2 | to | | L.,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | |
| | | Date | Time start | Time end | NMES intensity | Stretching | Notes |
| | 1.<br>2 | | | | | | |
| | 3 | | | | | | |
| | 4. | | | | | | |
| Outpatient therapy session: Yes/ No Date: Time: Fromto Place: | Dat<br>Tim | te:<br>ne: From | | | | | |

## Week 3

| No | Date | Time start | Time end | NMES intensity | Stretching | Notes |
|----|------|------------|----------|----------------|------------|-------|
| 1. | | | | | | |
| 2. | | | | | | |
| 3. | | | | | | |
| 4. | | | | | | |
| 5. | | | | | | |

| Da<br>Ti | ate: | apy session: Yes | | | | |
|---|---|---|---|---|---|---|
| W | <u>'eek 4</u> | | | | | |
| No | Date | Time start | Time end | NMES intensity | Stretching | Notes |
| 1. | | | | | | |
| 1.<br>2.<br>3.<br>4. | | | | | | |
| 3. | | | | | | |
| 4. | | | | | | |
| 5. | | | | | | |
| Da | ate: | apy session: Yes<br>to | | | | |
| | ace: | | | | | |